CLINICAL TRIAL: NCT01067716
Title: A Prospective Study to Evaluate the Performance and Acceptability of Advanced Variable Spot Scanning (AVSS) Ablations With the STAR S4 IR® Excimer Laser System
Brief Title: Performance and Acceptability of VSS-R
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Optics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STAR-107-AVSS
Record Dates: First submitted 2010-02-10; First posted 2010-02-12 (Estimated); Results first posted 2013-05-22 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2013-10

CONDITIONS: Refractive Error
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Refractive Error (Experimental)
  Interventions: Device: STAR S4IR LASIK with VSS-R ablation profile

INTERVENTIONS:
Device: STAR S4IR LASIK with VSS-R ablation profile — LASIK treatment targeted for emmetropia

SUMMARY:
The results of this trial will demonstrate that AVSS software performs as intended and is acceptable in a clinical setting.

DETAILED DESCRIPTION:
LASIK treatment across the range of myopia with or without astigmatism, hyperopia with or without astigmatism, and mixed astigmatism.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, of any race, and at least 21 years old at the time of the pre-operative examination and signing the consent form.
* The refractive error, based on manifest refraction at the spectacle plane, of: MRSE up to -15.00 D with manifest cylinder between 0.00 and -6.00 D; MRSE up to +7.00 D, with manifest cylinder between 0.00 and 6.00 D; or Manifest cylinder (from 1.0 to 6.0 D) greater than the magnitude of sphere, and the manifest cylinder and sphere have opposite signs.
* BSCVA of 20/20 or better.
* UCVA of 20/40 or worse.
* Manifest refraction sphere within ± 0.75 D of cycloplegic refraction sphere (at the same vertex distance).
* Anticipated post-operative stromal bed thickness of at least 250 microns, based on pre-operative central corneal pachymetry minus the maximum treatment depth to be ablated and the intended flap thickness, and confirmed by intra-operative central corneal pachymetry.
* Anticipated post-operative keratometry value (based on pre-operative manifest refraction and keratometry) that is appropriate.
* A stable refractive error, based on an exam (or prescription) at least 12 months prior to the pre-operative examination and as compared to the pre-operative manifest refraction
* Subjects who have worn a contact lens in the operative eye must discontinue lens wear at least three (3) consecutive weeks prior to the pre-operative examination. If, upon review of pre-operative measurements, the Investigator determines that the corneal topography is within normal limits, surgery may be scheduled (within 60 days), with no contact lens wear permitted prior to the surgery.
* Willing and capable of returning for follow-up examinations for the duration of the study (6 months).

Exclusion Criteria:

* Women who are pregnant, breast-feeding, or intend to become pregnant over the course of the study, as determined by verbal inquiry.
* Concurrent use of topical or systemic medications that may impair healing, including but not limited to: antimetabolites, isotretinoin (Accutane®) within 6 months of treatment, and amiodarone hydrochloride (Cordarone®) within 12 months of treatment.
* History of any of the following medical conditions, or any other condition that could affect wound healing: collagen vascular disease, autoimmune disease, immunodeficiency diseases, ocular herpes zoster or herpes simplex, endocrine disorders (including, but not limited to unstable thyroid disorders and diabetes), lupus, and rheumatoid arthritis.
* Subjects with a cardiac pacemaker or implanted defibrillator.
* History of prior intraocular or corneal surgery (including cataract extraction), active ophthalmic disease or abnormality (including, but not limited to, symptomatic blepharitis, recurrent corneal erosion, dry eye syndrome, neovascularization > 1mm from limbus), retinal detachment/repair, clinically significant lens opacity, clinical evidence of trauma, corneal opacity within the central 9 mm, at risk for developing strabismus, or with evidence of glaucoma or propensity for narrow angle glaucoma.
* Evidence of keratoconus, corneal dystrophy or irregularity, or abnormal videokeratography.
* Known sensitivity or inappropriate responsiveness to any of the medications used in the post-operative course.
* Subjects with one eye that does not meet all inclusion criteria and does not fall within approved indications for treatment using the VISX® STAR S4 IR® Excimer Laser.
* Participation in any other clinical study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2010-02; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Tarantino, OD, Study Director — Abbott Medical Optics
Locations (5):
- Canada (5):
  - Valley Laser Eye Centre, Abbottsford, British Columbia
  - Clearly LASIK, Victoria, British Columbia
  - Image Plus Laser Eye Center, Winnipeg, Manitoba
  - University of Ottawa Eye Institute, Ottawa, Ontario
  - Yonge-Eglington Laser, Toronto, Ontario

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One or both eyes of 79 subjects (150 eyes) were treated.
Groups:
- Myopia With and Without Astigmatism: Myopia with and without astigmatism with MRSE up to -15.0D, with cylinder between 0.00 and -6.00 D.
- Hyperopia With and Without Astigmatism: Hyperopia with and without astigmatism with MRSE up to +9.00 D, with cylinder between 0.00 and +6.00 D.
- Mixed Astigmatism: Mixed Astigmatism when the magnitude of cylinder (from 1.0 to 6.0D) is greater than the magnitude of sphere, and the cylinder and sphere have opposite signs.
Period: Overall Study
Arm/Group | Myopia With and Without Astigmatism | Hyperopia With and Without Astigmatism | Mixed Astigmatism
Started | 57 (110 eyes) | 13 (25 eyes) | 9 (15 eyes)
Completed | 57 (110 eyes) | 13 (25 eyes) | 9 (15 eyes)
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Myopia With or Without Astigmatism: Myopia with and without astigmatism with MRSE up to -15.0D, with cylinder between 0.00 and -6.00 D.
- Total: Total of all reporting groups
Arm/Group | Myopia With or Without Astigmatism | Hyperopia With and Without Astigmatism | Mixed Astigmatism | Total
Number analyzed (Participants) | 57 | 13 | 9 | 79
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 57 | 13 | 9 | 79
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 9 | 4 | 38
  Male | 32 | 4 | 5 | 41
Region of Enrollment [Number; unit: participants]
  Canada | 57 | 13 | 9 | 79

OUTCOME MEASURES:

1. Primary Outcome: Percent of Eyes With Uncorrected Visual Acuity (UCVA) of 20/40 or Better
Time Frame: 1 Year
Population: As a measure of effectiveness of LASIK treatment with VSS, distance visual performance without spectacles, clinically measured as Uncorrected Visual Acuity (UCVA) will be measured under standardized conditions such as 4 meter testing distance, controlled ambient room lighting and standard eye charts.
Measure: Number (95% Confidence Interval); unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Myopia With and Without Astigmatism | Hyperopia With and Without Astigmatism | Mixed Astigmatism
Number analyzed (Participants) | 57 | 13 | 9
Number analyzed (eyes) | 110 | 25 | 15
percentage of eyes | 99.1 [95.0 to 100.0] | 96.0 [79.6 to 99.9] | 100.0 [81.9 to 100.0]

2. Other Pre Specified Outcome: Percent Manifest Refraction Spherical Equivalent Within 1.0D
Description: Manifest refraction spherical equivalent is the required spectacle (or glass) prescription.
Time Frame: 1 Year
Population: As a measure of effectiveness of LASIK treatment with VSS, the required spectacle prescription, also called manifest refraction, will be measured under standardized conditions such as 4 meter testing distance, controlled ambient room lighting and standard eye charts.
Measure: Number (95% Confidence Interval); unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Myopia With and Without Astigmatism | Hyperopia With and Without Astigmatism | Mixed Astigmatism
Number analyzed (Participants) | 57 | 13 | 9
Number analyzed (eyes) | 110 | 25 | 15
percentage of eyes | 96.4 [91.0 to 99.0] | 92.0 [74.0 to 99.0] | 100.0 [81.9 to 100.0]

3. Other Pre Specified Outcome: Loss of More Than 2 Lines Best Spectacle Corrected Visual Acuity (BSCVA)
Description: After surgery, with or without best spectacle prescription the subject is not expected to see worse than before surgery. As a metric for this safety endpoint, losses of 2 lines of vision on a standard eye chart, with best spectacle correction, after surgery compared to pre-operative baseline shall be evaluated. For example 20/20 is typically considered best vision and 2 lines worse than this will be 20/32).
Time Frame: 1 Year
Measure: Number (95% Confidence Interval); unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Myopia With and Without Astigmatism | Hyperopia With and Without Astigmatism | Mixed Astigmatism
Number analyzed (Participants) | 57 | 13 | 9
Number analyzed (eyes) | 110 | 25 | 15
percentage of eyes | .9 [0.0 to 5.0] | 4.0 [0.1 to 20.4] | 0.0 [NA to NA] — Confidence intervals were not calculated because 0% of eyes had a loss of more than 2 lines of BSCVA

4. Other Pre Specified Outcome: Induced Manifest Refractive Astigmatism Greater Than 2.0 D of Absolute Cylinder Power
Time Frame: 1 Year
Measure: Number (95% Confidence Interval); unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Myopia With and Without Astigmatism | Hyperopia With and Without Astigmatism | Mixed Astigmatism
Number analyzed (Participants) | 57 | 13 | 9
Number analyzed (eyes) | 110 | 25 | 15
percentage of eyes | 0.0 [NA to NA] — Confidence intervals were not calculated because 0% of eyes had induced manifest refractive astigmatism greater than 2.0 D of absolute cylinder power. | 0.0 [NA to NA] — Confidence intervals were not calculated because 0% of eyes had induced manifest refractive astigmatism greater than 2.0 D of absolute cylinder power. | 0.0 [NA to NA] — Confidence intervals were not calculated because 0% of eyes had induced manifest refractive astigmatism greater than 2.0 D of absolute cylinder power.

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Myopia With or Without Astigmatism | Hyperopia With and Without Astigmatism | Mixed Astigmatism
Serious Adverse Events (participants affected / at risk) | 0/57 | 1/13 | 0/9
Other Adverse Events (participants affected / at risk) | 17/57 | 12/13 | 0/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Myopia With or Without Astigmatism (N=57) | Hyperopia With and Without Astigmatism (N=13) | Mixed Astigmatism (N=9)
Decrease in BSCVA of greater than or equal to two lines (Eye disorders) | 0 (0) | 1 (1) | 0 (0) — Loss of greater than or equal to two lines of BSCVA is an SAE in the context of this study.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Myopia With or Without Astigmatism (N=57) | Hyperopia With and Without Astigmatism (N=13) | Mixed Astigmatism (N=9)
Inadvertent insallation of Tropicamide instead of Tetracaine (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Elevated IOP (temporary) (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Photic phenomena (i.e., halos, glare, starbursts) (Eye disorders) | 9 (9) | 2 (2) | 0 (0)
Corneal Haze (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 4 (4) | 5 (5) | 0 (0)
Double vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Superficial epithelial linear laceration (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral infiltrates (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Other - hairline ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Other - cold/flu (General disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At least ninety (90) days prior to any proposed submission for publication or presentation of Study Data or other findings related to the Study, Institution will provide Sponsor with a manuscript of such submission(s) for review, comment, and approval. For greater certainty, neither Institution nor Principal Investigator shall have any right to publish any information or results concerning the Study without the express written consent of Sponsor.